CLINICAL TRIAL: NCT04206124
Title: Regulation of Beige Fat Development by mTORC1 and Autophagy
Brief Title: mTORC1 and Autophagy in Human Brown Adipocytes
Acronym: mTORHBFC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Meilian Liu, Associate Professor, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-272
Record Dates: First submitted 2019-12-13; First posted 2019-12-20 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Obesity; Metabolic Disease
Keywords: Autophagy; Inflammation; Metabolism; Adipocyte; mTORC1; Obesity; Thermogenesis
MeSH Terms: conditions — Obesity; Metabolic Diseases; Inflammation

STUDY DESIGN:
Intervention Model Description: Patients will be recruited based on sex, age, and medical history including BMI (lean, <25, or obese, >30), medication list, and health status. Included patients indicated for thyroidectomy, parathyroidectomy, or cervical spine injury surgery, who are able to consent, will have a soybean-sized amount of brown fat removed from the neck during surgery. These tissue samples will be further analyzed using biochemical tools after being de-identified from patient records.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Study Group (Experimental): Includes all consented patients, male and female, undergoing anterior cervical spine surgery, parathyroidectomy or thyroidectomy (18-60 years old), without history of diabetes mellitus and not pregnant or incarcerated.
  Interventions: Procedure: Brown Fat Harvest During Anterior Neck Surgery

INTERVENTIONS:
Procedure: Brown Fat Harvest During Anterior Neck Surgery — During previously indicated thyroid gland removal or anterior cervical spine surgery, as scheduled at UNMHSC, the surgeon will identify the large muscle on the side of the neck in the surgical field. Using minimal dissection adjacent to the muscle, they will then remove 5-10mg of brown fat from this region. These samples will be further analyzed using various biochemical tools.

SUMMARY:
The long term goal is to identify the potential therapeutic targets for the treatment of obesity and its associated disorders by studying the driving factors of activation of brown adipose tissue (BAT) in human adults. Whereas activation of brown adipose tissue (BAT) in human adults has been considered as a potential therapeutic target to battle obesity since it was identified in 2009, the underlying mechanisms of beige adipocytes appearance in human adults is unclear. The objective of this proposal is to investigate the role of autophagy in mediating the inhibitory effect of mammalian target of rapamycin complex 1 (mTORC1) in regulating human brown adipocytes. The central hypothesis is that autophagy plays a critical role in regulating browning of white adipose tissue and mediates the beneficial effect of mTORC1 inhibition on thermogenesis in human brown adipocytes.

DETAILED DESCRIPTION:
Specific Aim 1: To investigate the role of mTORC1 and autophagy in regulating thermogenesis in human brown adipocytes. The working hypothesis is that inhibition of mTORC1 or activation of autophagy improves thermogenesis in human brown adipocytes. It will be first determined if the mTORC1/autophagy signaling modulates thermogenic gene expression and beige markers by collecting human brown fat from lean non-diabetic subjects. The brown fat during the anterior cervical spine surgery or thyroidectomy from lean subjects with a BMI <25, or obese participants who have a BMI >30, will be harvested and then be used to determine: 1) whether mTORC1 signaling, autophagy and thermogenic gene expression, and the fraction of various types of immune cells in human brown fat are different from those in rodents;2) whether rapamycin treatment enhances basal or CL-induced thermogenic gene expression and O2 consumption in primary human brown adipocytes; and 3) whether inhibition of autophagy by 3-methyladenine (3-MA) suppresses thermogenic gene expression induced by CL316,243, a β3-adrenoceptor agonist that mimics cold stress in vivo in human brown adipocytes.

Overall, this study will lead to the identification of mTORC1 as a key regulator of thermogenesis in human adipose tissue and reveal promising new anti-obesity drug targets. In addition, this study will further investigate the role of rapamycin administration in obesity in human adults near the future. These studies are designed to be a proof-of-principle. If the results are promising, then future drug development could focus on designing new inhibitors of mTORC1.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* age 18-60
* able to give informed consent
* non-diabetic
* scheduled for anterior cervical spine, thyroidectomy, or parathyroidectomy surgery at UNMHSC
* BMI <25 (lean) or >30 (obese)
* English or Spanish speaking

Exclusion Criteria:

* has diabetes mellitus (type I or II)
* currently on any study medication (including sedatives or analgesics, coagulopathy (INR of 1.5 or greater, platelet count of <50,000/microliter), or anticoagulant)
* pregnant
* incarcerated

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Protein expression levels in lean and obese human brown adipose tissue samples will be quantified via Western Blot and comparatively analyzed using a student T-test. | Up to six years after date of sample collection.
  Human brown adipose tissue (BAT) samples will be collected during previously scheduled anterior neck surgery and then cultured and amplified for experiments including Western Blot (WB), an assay to quantify the relative amounts of protein present in a sample.
  WB will be used to determine how protein expression levels differ between lean and obese BAT samples. Specifically, the translational levels of key markers of mTOR signaling including UCP1, C/EBPβ, HSL, S6K, ADPN, PKA, AMPK and ATGL will be quantified by WB and analyzed statistically using student T-test, and protein activation levels will be quantified by dividing phosphorylated protein content by total protein content.
Gene transcript expression levels in lean and obese human brown adipose tissue samples will be quantified via quantitative Polymerase Chain Reaction and comparatively analyzed using a student T-test. | Up to six years after date of sample collection.
  Human brown adipose tissue (BAT) samples will be collected during previously scheduled anterior neck surgery and then cultured and amplified for experiments including quantitative-Polymerase Chain Reaction (q-PCR), an assay to quantify the relative amounts of mRNA (transcribed genes) present in a sample.
  q-PCR will be used to determine how gene expression levels differ between lean and obese BAT samples. Specifically, the transcriptional levels of key markers of mTOR signaling including UCP1, C/EBPβ, HSL, S6K, ADPN, PKA, AMPK and ATGL will be quantified by q-PCR and analyzed using student T-test.

CONTACTS AND LOCATIONS:
Overall Officials: Meilian Liu, PhD, Principal Investigator — University of New Mexico Biochemistry & Molecular Biology
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will be de-identified after specimen collection. De-identified data will be stored securely and not shared with other researchers.